CLINICAL TRIAL: NCT00657189
Title: A Phase 2A , Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Dose Study to Evaluate the Safety and Tolerability of Multiple Subcutaneous Doses of MEDI-545, A Fully Human Anti-Interferon-Alpha Monoclonal Antibody, In Subjects With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate Safety and Tolerability of Subcutaneous Doses of MEDI-545 in Subjects With Lupus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP179
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Lupus Erythematosus, Systemic; Lupus
Keywords: Sifalimumab; MEDI-545; Lupus erythematosus, systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — sifalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): MEDI-545
  Interventions: Drug: MEDI-545
- 2 (Experimental): MEDI-545
  Interventions: Drug: MEDI-545
- 3 (Experimental): MEDI-545
  Interventions: Drug: MEDI-545
- 4 (Experimental): MEDI-545
  Interventions: Drug: MEDI-545
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI-545 — 100 mg once; SC Placebo × 12 doses on other weeks
  Arms: 1
Drug: MEDI-545 — 100 mg every 4 weeks × 4 doses; SC Placebo × 9 doses on other weeks
  Arms: 2
Drug: MEDI-545 — 100 mg every 2 weeks × 7 doses; SC Placebo × 6 doses on other weeks
  Arms: 3
Drug: MEDI-545 — 100 mg every week × 13 doses
  Arms: 4
Drug: Placebo — SC Placebo every week × 13 doses
  Arms: 5

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of multiple doses of MEDI-545 in subjects with moderately to severely active Lupus.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of multiple SC doses of MEDI-545 in subjects ≥ 18 years of age with moderately to severely active SLE despite standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years at the time of the first dose of study drug;
* Written informed consent and HIPAA authorization (applies to covered entities in the US only) obtained from the subject or subject's legal representative;
* Meet at least 4 of the 11 revised ACR classification criteria for SLE
* Have positive antinuclear antibody test (ANA) at ≥ 1:80 serum dilution documented in the past or at screening;
* Have at least 1 system with a score of A or 2 systems with a score of B on the BILAG index at screening, or have a SELENA-SLEDAI score ≥ 6;
* Treatment for SLE with antimalarials, oral prednisone or another systemic corticosteroid, mycophenolate mofetil, methotrexate, leflunomide, azathioprine, or dapsone;
* Women, unless surgically sterile or at least 2 years post-menopausal, must use an effective method of avoiding pregnancy (including oral, injectable, transdermal, or implanted contraceptives, intrauterine device, diaphragm with spermicide, cervical cap, abstinence, or sterile sexual partner) in addition to the use of condoms (male or female condoms with spermicide) from screening through the end of the study. Cessation of birth control after this point should be discussed with a responsible physician. Men unless surgically sterile, must likewise practice 2 effective methods of birth control (condom with spermicide or abstinence) from Study Day 0 through the end of the study;
* Ability to complete the study period, including the follow-up period through Study Day 168; and
* Willing to forego other forms of experimental treatment during the study.

Exclusion Criteria:

* Have received MEDI-545 within 120 days prior to screening;
* History of allergy or reaction to any component of the study drug formulation;
* Have received the following medications within 28 days before randomization:

  * Systemic cyclophosphamide at any dose
  * Cyclosporine at any dose
  * Thalidomide at any dose
  * Hydroxychloroquine > 600 mg/day
  * Mycophenolate mofetil > 3 g/day
  * Methotrexate > 25 mg/week
  * Azathioprine > 3 mg/kg/day
* Have received fluctuating doses of the following within 28 days before randomization:

  * Antimalarials
  * Mycophenolate mofetil
  * Methotrexate
  * Leflunomide
  * Azathioprine
  * Dapsone
* Have received Leflunomide > 20mg/day in the 6 months prior to Study Day 0;
* Have received prednisone > 20 mg/day or in fluctuating doses within 14 days before randomization;
* Have received fluctuating doses of non-steroidal anti-inflammatory drugs within 14 days before randomization;
* Treatment with any investigational drug therapy within 28 days before randomization into the study, B cell-depleting therapies within 12 months before randomization, or biologic therapies within 30 days or 5 half-lives of the biologic agent, whichever is longer, before randomization into the study;
* In the investigator's opinion, evidence of clinically significant active infection, including ongoing, chronic infection, within 28 days before randomization;
* A history of severe viral infection as judged by the investigators, including severe infections of either cytomegalovirus or the herpes family such as disseminated herpes, herpes encephalitis, ophthalmic herpes;
* Herpes zoster infection within 3 months before randomization;
* Evidence of infection with hepatitis B or C virus, or human immunodeficiency virus (HIV)-1 or HIV-2, or active infection with hepatitis A, as determined by results of testing at screening
* Vaccination with live attenuated viruses within 28 days before randomization;
* Pregnancy (women, unless surgically sterile or at least 2 years post-menopausal, must have a negative serum pregnancy test within 28 days before receiving the study drug and a negative urine pregnancy test on days of study drug administration before receiving the study drug);
* Breastfeeding or lactating women;
* History of primary immunodeficiency;
* History of alcohol or drug abuse < 1 year prior to randomization;
* History of cancer (except basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy > 1 year prior to randomization);
* History of active tuberculosis (TB) infection or newly positive TB skin test (defined as a reaction ≥ 10 mm in diameter if not on systemic immunosuppressive medication or ≥ 5 mm if on systemic immunosuppressive medication;
* History of latent TB infection without completion of an appropriate course of treatment;
* Elective surgery planned from the time of screening through Study Day 168;
* At screening blood tests (within 28 days before randomization), any of the following:

  * AST > 2.5 x upper limit of the normal range (ULN), unless caused by SLE
  * ALT > 2.5 x ULN, unless caused by SLE
  * Creatinine > 4.0 mg/dL
  * Neutrophils < 1,500/mm3
  * Platelet count < 50,000/mm3
* History of any disease, evidence of any current disease (other than SLE), any finding upon physical examination, or any laboratory abnormality that, in the opinion of the investigator or medical monitor, may compromise the safety of the subject in the study or confound the analysis of the study; or
* Any employee of the research site who is involved with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of MEDI-545 will be assessed primarily by summarizing treatment emergent AEs and SAEs and by assessing changes in viral cultures. | Immediately following the first administration of study drug through Study Day 168.

SECONDARY OUTCOMES:
A secondary endpoint of this study is to assess certain measures of disease activity including PK, and PD of SC doses of MEDI-545. | At Study Day 98

CONTACTS AND LOCATIONS:
Overall Officials: Warren Greth, M.D., Study Director — MedImmune LLC
Locations (22):
- United States (22):
  - Research Site, Anniston, Alabama
  - Research Site, Huntington Beach, California
  - Research Site, Upland, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Farmington, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Ocala, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Marrietta, Georgia
  - Research Site, West Fayetteville, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Lansing, Michigan
  - Research Site, Brooklyn, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Houston, Texas
  - Research Site, Sugarland, Texas
  - Research Site, Seattle, Washington

REFERENCES:
- [Result] Merrill JT, Wallace DJ, Petri M, Kirou KA, Yao Y, White WI, Robbie G, Levin R, Berney SM, Chindalore V, Olsen N, Richman L, Le C, Jallal B, White B; Lupus Interferon Skin Activity (LISA) Study Investigators. Safety profile and clinical activity of sifalimumab, a fully human anti-interferon alpha monoclonal antibody, in systemic lupus erythematosus: a phase I, multicentre, double-blind randomised study. Ann Rheum Dis. 2011 Nov;70(11):1905-13. doi: 10.1136/ard.2010.144485. Epub 2011 Jul 27. PMID 21798883